CLINICAL TRIAL: NCT02638207
Title: Prospective, Double-blind, Randomized, Multicenter Phase III Study Evaluating Efficacy and Safety of Three Different Dosages of NewGam in Patients With Chronic Inflammatory Demyelinating Poly(Radiculo)Neuropathy
Brief Title: Study to Evaluate Safety and Efficacy of Three Different Dosages of NewGam in Patients With Chronic Inflammatory Demyelinating Poly (Radiculo) Neuropathy
Acronym: CIDP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGAM-08
Record Dates: First submitted 2015-12-16; First posted 2015-12-23 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Chronic Inflammatory Demyelinating Poly(Radiculo)Neuropathy
Keywords: Chronic Inflammatory Demyelinating Poly Neuropathy (CIDP)
MeSH Terms: interventions — Panzyga

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.5 g/kg NewGam (Experimental): All patients will receive a loading dose of 2.0 g/kg Newgam (administered over two consecutive days), followed by seven infusions of the maintenance dose the patient has been randomized to (0.5g/kg NewGam), also administered over two consecutive days every 3 weeks (±4 days).
  Interventions: Drug: NewGam
- 1.0 g/kg NewGam (Experimental): All patients will receive a loading dose of 2.0 g/kg Newgam (administered over two consecutive days), followed by seven infusions of the maintenance dose the patient has been randomized to (1.0g/kg NewGam), also administered over two consecutive days every 3 weeks (±4 days).
  Interventions: Drug: NewGam
- 2.0 g/kg NewGam (Experimental): All patients will receive a loading dose of 2.0 g/kg Newgam (administered over two consecutive days), followed by seven infusions of the maintenance dose the patient has been randomized to (2.0g/kg NewGam), also administered over two consecutive days every 3 weeks (±4 days).
  Interventions: Drug: NewGam

INTERVENTIONS:
Drug: NewGam — In the Dose-evaluation Phase, all patients will receive a loading dose of 2.0 g/kg Newgam (administered over two consecutive days), followed by seven infusions of the maintenance dose the patient has been randomized to (0.5, 1.0 or 2.0 g/kg NewGam), also administered over two consecutive days every 3 weeks (±4 days). If a patient is randomized to receive the low or medium NewGam dose, the same volume with the same infusion rate as would have been applied in case the patient would have been randomized to 2.0 g/kg NewGam will be used, thus supplemented with an authorized 0.9% w/v isotonic sodium chloride solution as appropriate and detailed in the following infusion bag split to maintain the blinding
  Other Names: Panzyga

SUMMARY:
Study to evaluate the Efficacy and Safety of Three Different Dosages of NewGam in Patients With Chronic Inflammatory Demyelinating Poly(radiculo)neuropathy

DETAILED DESCRIPTION:
Prospective, Double-blind, Randomized, Multicenter Phase III Study Evaluating Efficacy and Safety of Three Different Dosages of NewGam in Patients With Chronic Inflammatory Demyelinating Poly(radiculo)neuropathy ("ProCID trial")

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of definite or probable Chronic inflammatory demyelinating polyneuropathy (CIDP) according to the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) Guideline 2010 [van den Bergh et al., 2010]; including patients with Multifocal Acquired Demyelinating Sensory And Motor Neuropathy (MADSAM) or pure motor Chronic inflammatory demyelinating polyneuropathy (CIDP )
2. Patients currently depending on treatment with immunoglobulins or corticosteroids
3. Patients with active disease, i.e. not being in remission, who are progressive or relapsing prior to trial start or during the Wash-out Phase
4. Weakness of at least 2 limbs
5. >18 to <80 years of age
6. Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score between 2 and 9 (with a score of 2 coming exclusively from leg disability)
7. Voluntarily given, fully informed written consent obtained from patient before any study-related procedures are conducted

Exclusion Criteria:

1. Unifocal forms of Chronic inflammatory demyelinating polyneuropathy (CIDP)
2. Pure sensory Chronic inflammatory demyelinating polyneuropathy (CIDP)
3. Multifocal motor neuropathy (MMN) with conduction block [van den Bergh et al., 2010]
4. Patients who previously failed immunoglobulin treatment
5. Treatment with immunomodulatory/suppressive agents (cyclosporin, methotrexate, mitoxantrone, mycophenolate mofetil or azathioprine) during the six months prior to baseline visit
6. Patients on or treated with rituximab, alemtuzumab, cyclophosphamide, or other intensive chemotherapeutic regimens, previous lymphoid irradiation or stem cell transplantation during the 12 months prior to baseline visit
7. Respiratory impairment requiring mechanical ventilation
8. Myelopathy or evidence of central nervous system demyelination or significant persisting neurological deficits from stroke, or central nervous system (CNS) trauma
9. Clinical evidence of peripheral neuropathy from another cause such as

   1. connective tissue disease or systemic lupus erythematosus (SLE)
   2. HIV infection, hepatitis, Lyme disease
   3. cancer (with the exception of basal cell skin cancer)
   4. IgM paraproteinemia with anti-myelin associated glycoprotein antibodies
10. Diabetic neuropathy
11. Cardiac insufficiency (New York Heart Association [NYHA] III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease
12. Severe liver disease (ALAT 3x > normal value)
13. Severe kidney disease (creatinine 1.5x > normal value)
14. Hepatitis B, hepatitis C or HIV infection
15. Thromboembolic events: patients with a history of deep vein thrombosis (DVT) within the last year prior to baseline visit or pulmonary embolism ever; patients with susceptibility to embolism or deep vein thrombosis (DVT)
16. Body mass index (BMI) ≥40 kg/m2
17. Patients with uncompensated hypothyroidism (abnormally high Thyroid-Stimulating Hormone [TSH] and abnormally low Thyroxine [T4]) or known vitamin B12 deficiency if patients don't receive adequate substitution therapy
18. Medical conditions whose symptoms and effects could alter protein catabolism and/or Immunoglobulin G (IgG) utilization (e.g. protein-losing enteropathies, nephrotic syndrome)
19. Known Immunoglobulin A (IgA) deficiency with antibodies to Immunoglobulin A (IgA)
20. History of severe hypersensitivity, e.g. anaphylaxis or severe systemic response to immuno-globulin, blood or plasma derived products, or any component of NewGam
21. Known blood hyperviscosity, or other hypercoagulable states
22. Use of other blood or plasma-derived products within three months prior to Visit 2
23. Patients with a past or present history of drug abuse or alcohol abuse within the preceding five years prior to baseline visit
24. Patients unable or unwilling to understand or comply with the study protocol
25. Participation in another interventional clinical study with investigational medicinal product (IMP) treatment currently or during the three months prior to Visit 2
26. Women who are breast feeding, pregnant, or planning to become pregnant, or are unwilling to use an effective birth control method (such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner) while on study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, MD, Study Director — Octapharma
Locations (26):
- Bulgaria (2):
  - MHAT Puls EOOD, Blagoevgrad
  - St. Naum Hospital, Sofia
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Octapharma Research Site, Montreal
- Czechia (3):
  - Outpatient Clinic of Neurology, Hradec Králové
  - Regional Hospital Pardubice, Pardubice
  - Thomayer Faculty Hospital, Prague
- University Medical Center Goettigen, Goettigen, Germany
- Hungary (2):
  - Jahn Ferenc Del Pesti Korhaz, Budapest
  - Szegedi Tudományegyetem ÁOK Neurológiai Klinika, Szeged
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie Klinika Neurologii, Lublin
  - Wojewodzki Szpital Specjalistyczny W Olsztynie, Olsztyn
  - Uniwersytecki Szpital Kliniczny, Wroclaw
- Romania (3):
  - Theo Health S.R.L., Brasov
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Judetean de Urgenta "Sf.Apostol Andrei" Constanta, Constanța
- Russia (5):
  - Republican Clinical Neurological Centre, Kazan'
  - Neurology Research Centre, Moscow
  - Nizhny Novgorod Regional Clinical Hospital N.A. N.A.Semashko, Nizhny Novgorod
  - National Medical Research Centre of Psychiatry and Neurology n.a. V.M.Bekhterev, Saint Petersburg
  - City Multifield Hospital #2, Saint Petersburg
- Ukraine (5):
  - Ivano Frankivsk National Medical University, Ivano-Frankivsk
  - National Medical Academy Of Postgraduate Education Named After P.L. Shupyk, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Vinnytsia National Medical University, Vinnytsia
  - Municipal Institution Zaporizhzhya Regional Clinical Hospital, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bus SR, de Haan RJ, Vermeulen M, van Schaik IN, Eftimov F. Intravenous immunoglobulin for chronic inflammatory demyelinating polyradiculoneuropathy. Cochrane Database Syst Rev. 2024 Feb 14;2(2):CD001797. doi: 10.1002/14651858.CD001797.pub4. PMID 38353301
- [Derived] Cornblath DR, van Doorn PA, Hartung HP, Merkies ISJ, Katzberg HD, Hinterberger D, Clodi E; ProCID Investigators. Safety and Tolerability of Intravenous Immunoglobulin in Chronic Inflammatory Demyelinating Polyneuropathy: Results of the ProCID Study. Drug Saf. 2023 Sep;46(9):835-845. doi: 10.1007/s40264-023-01326-z. Epub 2023 Jun 28. PMID 37378806
- [Derived] Cornblath DR, van Doorn PA, Hartung HP, Merkies ISJ, Katzberg HD, Hinterberger D, Clodi E; ProCID Investigators. Randomized trial of three IVIg doses for treating chronic inflammatory demyelinating polyneuropathy. Brain. 2022 Apr 29;145(3):887-896. doi: 10.1093/brain/awab422. PMID 35038723

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Started | 35 | 69 | 38
Completed | 28 | 61 | 34
Not Completed | 7 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam | Total
Number analyzed (Participants) | 35 | 69 | 38 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.49 (14.449) | 56.32 (14.616) | 58.05 (13.764) | 55.84 (14.398)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 31 | 14 | 58
  Male | 22 | 38 | 24 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 35 | 69 | 38 | 142
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 84.09 (16.511) | 81.74 (16.333) | 77.68 (75.50) | 81.23 (79.00)
Height [Mean (Standard Deviation); unit: cm] | 173.46 (9.506) | 172.81 (8.304) | 171.61 (9.030) | 172.65 (8.770)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.92 (4.873) | 27.27 (4.588) | 26.33 (5.231) | 27.18 (4.837)

OUTCOME MEASURES:

1. Primary Outcome: Decrease in the Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Score
Description: Efficacy - Proportion of responders in the 1.0 g/kg NewGam arm at Week 24 (Termination Visit) relative to baseline (Week 0). A responder being defined as a patient with a decrease of at least 1 point on the adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score (a scale from 0 to 10, from healthy to unable to make any purposeful movements with arms and/or legs)
Time Frame: at Week 24
Population: Intention-to-treat Set (ITTS): The ITTS consist of all patients of the Safety Data Set for whom any data was collected post infusion of IMP. Three patients (one in the 0.5 g/kg group and two in the 2.0 g/kg group) were excluded from the ITTS as no data were collected post-infusion of IMP. Therefore n=139 for the ITTS. Every treated subject will be considered in the analysis according to his randomized treatment/dose assignment.
Measure: Number; unit: proportion of subjects
Arm/Group | 1.0 g/kg NewGam
Number analyzed (Participants) | 69
proportion of subjects | .7971

2. Secondary Outcome: Decrease in the Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Score
Description: Proportion of responders in the 0.5 g/kg and 2.0 g/kg NewGam arms at Week 24 relative to baseline compared to the 1.0 g/kg arm, based on the adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score
Time Frame: at Week 24
Population: as for outcome 1
Measure: Number; unit: Proportion of responders
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
Proportion of responders | .6471 | .7971 | .9167

3. Secondary Outcome: Grip Strength Score
Description: Proportion of responders in the 0.5 g/kg and 2.0 g/kg NewGam arms at Week 24 relative to baseline at Week 0 compared to the 1.0 g/kg arm, based on the grip strength (Martin Vigorimeter) using the previously published minimum clinically important difference (MCID) cut-off of 8 kilopascal (kPa)
Time Frame: at Week 24
Population: as for outcome 1
Measure: Number; unit: Proportion of responders
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
Proportion of responders | .5588 | .6522 | .8333

4. Secondary Outcome: Inflammatory Rasch-built Overall Disability Scale (I-RODS Score)
Description: Proportion of responders in the 0.5 g/kg and 2.0 g/kg NewGam arms at Week 24 relative to baseline at Week 0 compared to the 1.0 g/kg arm, based on the Inflammatory Rasch-built overall disability scale (I-RODS Score) using the MCID concept related to the varying standard errors (MCID-SE) as recently demonstrated
Time Frame: at Week 24
Population: as for outcome 1
Measure: Number; unit: Proportion of responders
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
Proportion of responders | .3824 | .5507 | .7222

5. Secondary Outcome: Worsening in the Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Score
Description: Time to first confirmed worsening on the adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability scale by at least 1 point from the value at baseline (Week 0)
Time Frame: Week 24
Population: There was only 1 patient with worsening (in the 1.0 g/kg group), thus an analysis of the time to first worsening was not possible.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
days | NA [NA to NA] — No patients with worsening in this group, analysis not possible. | NA [NA to NA] — There was only 1 patient with worsening (in the 1.0 g/kg group), thus an analysis of the time to first worsening was not possible. | NA [NA to NA] — No patients with worsening in this group, analysis not possible.

6. Secondary Outcome: Mean Change in Grip Strength
Description: Mean change from baseline (Week 0) to Termination Visit in grip strength of both hands (assessed by Martin vigorimeter). The reported change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
kPa
  Dominant Hand | 23.91 (25.290) | 19.38 (20.377) | 26.06 (25.030)
  Non-dominant Hand | 23.94 (24.600) | 17.43 (19.916) | 24.53 (22.247)

7. Secondary Outcome: Inflammatory Rasch-built Overall Disability Scale (I-RODS)
Description: Mean change from baseline (Week 0) to Termination Visit in Inflammatory Rasch-built overall disability sum score (I-RODS using the concept of MCID-SE as recently reported) and number of improvers. The reported change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
  A scale from 0 to 48, from "Not possible to perform" to "Possible without any difficulty". Higher values represent a better outcome.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
score on a scale | 11.38 (12.485) | 10.32 (10.836) | 13.86 (11.981)

8. Secondary Outcome: Motor Nerves
Description: Mean change from baseline (Week 0) to Termination Visit in sum of the distal evoked amplitude of 4 right sided and 4 left sided motor nerves (peroneal, tibial, ulnar and median). The reported change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 68 | 36
mV | 2.16 (6.332) | 2.69 (6.688) | 3.93 (9.298)

9. Secondary Outcome: Mean Change in Pain Intensity Numerical Rating Scale (PI-NRS Scale)
Description: Mean change from baseline (Week 0) to Termination Visit in Pain Intensity Numeric Rating Scale (PI-NRS). The reported change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
  The Pain Intensity Numeric Rating Scale (PI-NRS, a numeric scale where 0 = no pain and 10 = worst possible pain) is an 11-point scale for patient self-reporting of pain. A higher value represents a worse outcome.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
score on a scale | -2.29 (3.040) | -2.19 (2.907) | -2.17 (3.256)

10. Secondary Outcome: Worsening on the Inflammatory Rasch-built Overall Disability Scale (I-RODS Scale)
Description: Time to first confirmed worsening on the I-RODS scale. The reported change was calculated from two time points as the value at the later time point minus the value at the earlier time point. A scale from 0 to 48, from "Not possible to perform" to "Possible without any difficulty". Higher values represent a better outcome.
  Worsening is determined using the concept of MCID (minimum clinically important difference) using the individually obtained standard errors (MCID-SE).
Time Frame: 24 weeks
Population: There was 1 patient with worsening in the 0.5 g/kg group and 2 in the 1.0 g/kg group; an analysis of the time to first worsening was not possible
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
days | NA [NA to NA] — There was only 1 patient with worsening in this group, thus an analysis of the time to first worsening was not possible. | NA [NA to NA] — There were only 2 patients with worsening in this group, thus an analysis of the time to first worsening was not possible. | NA [NA to NA] — No patients with worsening in this group, analysis not possible.

11. Secondary Outcome: 1 Point Decrease in the INCAT Disability Score
Description: Time to 1 point decrease (improvement of disability) in adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
days | 22.0 [22.0 to 24.0] | 26.0 [22.0 to 43.0] | 23.0 [22.0 to 43.0]

12. Secondary Outcome: Decrease in Inflammatory Rasch-built Overall Disability Scale (I-RODS Scale)
Description: Time to decrease in Inflammatory Rasch-built overall disability scale (I-RODS) scores
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 0.5 g/kg NewGam | 1.0 g/kg NewGam | 2.0 g/kg NewGam
Number analyzed (Participants) | 34 | 69 | 36
days | NA [NA to NA] — There were no patients with worsening in this group thus an analysis of the time to first worsening was not possible. | NA [NA to NA] — There was only 1 patient with worsening in this group thus an analysis of the time to first worsening was not possible. | NA [NA to NA] — There were no patients with worsening in this group thus an analysis of the time to first worsening was not possible.

ADVERSE EVENTS:
Time Frame: Up to 36 weeks
Description: An AE is any untoward medical occurrence in a patient receiving an IMP and which does not have to have a causal relationship with treatment.
  At each visit AEs will be elicited using a standard non-leading question like "How have you been since the last visit / during the previous study period?" Patient diaries will also be checked.
  Safety Data Set (SDS): The SDS was based on all randomized patients who received at least part of one infusion of IMP. Therefore n=142 for the SDS.
Groups:
- NGAM 0.5 g/kg: NGAM 0.5 g/kg
- NGAM 1.0 g/kg: NGAM 1.0 g/kg
- NGAM 2.0 g/kg: NGAM 2.0 g/kg
- Total: Total of all three treatment arms.
Arm/Group | NGAM 0.5 g/kg | NGAM 1.0 g/kg | NGAM 2.0 g/kg | Total
All-Cause Mortality (participants affected / at risk) | 0/35 | 1/69 | 1/38 | 2/142
Serious Adverse Events (participants affected / at risk) | 1/35 | 4/69 | 1/38 | 6/142
Other Adverse Events (participants affected / at risk) | 20/35 | 45/69 | 24/38 | 88/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NGAM 0.5 g/kg (N=35) | NGAM 1.0 g/kg (N=69) | NGAM 2.0 g/kg (N=38) | Total (N=142)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardio-respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NGAM 0.5 g/kg (N=35) | NGAM 1.0 g/kg (N=69) | NGAM 2.0 g/kg (N=38) | Total (N=142)
Pyrexia (General disorders) | 3 (4) | 6 (6) | 2 (3) | 11 (13)
Chills (General disorders) | 3 (4) | 3 (3) | 1 (1) | 7 (8)
Influenza like illness (General disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Infusion site coldness (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Infusion site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 3 (7) | 6 (7) | 0 (0) | 9 (14)
Body temperature increased (Investigations) | 2 (2) | 4 (7) | 3 (3) | 9 (12)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 5 (5) | 0 (0) | 5 (5)
Heart rate decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Transaminases increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 9 (11) | 8 (12) | 19 (25)
Somnolence (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Tension headache (Nervous system disorders) | 0 (0) | 1 (4) | 1 (3) | 2 (7)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (10) | 4 (5) | 13 (19)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 4 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (5) | 2 (6)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Decubitis ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Eczema infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 3 (5) | 5 (8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 5 (5) | 0 (0) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (2) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (2) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (4) | 1 (1) | 4 (6)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Left atrial dilatation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (4)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gallbladder disorders (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctival oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT02638207/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT02638207/SAP_001.pdf